CLINICAL TRIAL: NCT03491722
Title: Evolution of Risk Factors and Revascularization Among >1 Decade Survivors After Coronary Revascularization in the Middle East
Brief Title: Surviving a Decade or More After Coronary Revascularization in a Middle Eastern Population
Acronym: DECADE1+ME
Status: Completed | Type: Observational
Sponsor: Jordan Collaborating Cardiology Group (Other)
Responsible Party: Principal Investigator, Ayman J Hammoudeh, MD, FACC, Interventional Cardiologist, Istishari Hospital, Amman, Jordan Collaborating Cardiology Group
Other Study IDs: DecadeOrMoreSurvivors01
Record Dates: First submitted 2018-04-02; First posted 2018-04-09 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Risk Factors AND Repeat Revascularization
MeSH Terms: interventions — Risk Factors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: risk factors and revascularization procedures — arterial revascularizations needed since index procedure

SUMMARY:
The study will look at the cardiovascular risk factors as they arise, as well at the need for further revascularization after at least 10 years of coronary revascularization in Middle Eastern patients.

The PI will overlook the whole process. Dr Ahmad Tamari, the assistant to the PI will asses this whole process of data collection, management and manuscript drafting.

DETAILED DESCRIPTION:
Middle Eastern patients aged 18 years or above presenting to cardiology service at one tertiary care center who had coronary revascularization (stent or coronary bypass surgery, i.e., index procedure) at least 10 years back, will interviewed to determine:

1. Evolution of cardiovascular risk factors in the period from index procedure to time of interview. These risk factors include; hypertension, diabetes, smoking, dyslipidemia and obesity.
2. Need for further arterial revascularization from the index procedure to time of interview.

   These arterial revascularization procedures include A. Coronary: stent and/or bypass surgery B. Carotid endarterectomy. C. peripheral arterial revascularization D. Renal artery stent.
3. Medications used at the time if interview with special emphases on the guideline-recommended medications including antiplatelet agents, beta blockers, statins and renin angiotensin blockers.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Coronary stent or bypass 10 years ago or more.
3. Dependable mental status to recall events.

Exclusion Criteria:

1. Non coronary operations
2. Inability to recall evnets

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All comers who had undergone coronary stent or bypass surgery 10 years or more prior to interview. These patients will be asked about the appearance of new cardiovascular risk factors during this period and whether they had undergone further operations or procedures to the coronary arteries, carotid arteries, lower limb arteries ir renal arteries.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Risk factors | Since index procedure to time of interview at least 10 years later
  Appearance of diabetes, hypertension, smoking, dyslipidemia or obesity since index procedure
Arterial revascularizations | Since index procedure to time of interview at least 10 years later
  Undergoing further coronary stent or surgery, carotid stent or surgery, lower limbs stent or surgery, and renal artery stent.

CONTACTS AND LOCATIONS:
Locations (2):
- Jordan (2):
  - Istishari Hospital, Amman
  - Specialty Hospital, Amman